CLINICAL TRIAL: NCT05217043
Title: Language Acquisition in the Brain and Algorithms: Towards Systematic Monitoring of the Evolution of Semantic Representations in Biological and Artificial Neural Networks
Acronym: SYNTAXE
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: PBN_2021_25
Record Dates: First submitted 2022-01-19; First posted 2022-02-01 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Language Acquisition in the Brain
Keywords: Intracranial recordings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: intracranial brain recording — Any patient benefiting from a long-term intracranial brain recording.

SUMMARY:
Speech depends on our ability to recursively combine successive words into a complex sense. Although the order of these putative operations (syntax) has been the subject of extensive examination in the way in which the human brain learns to perform a "Semantic composition" remains largely unknown.

The Rothschild Hospital houses a unit specializing in drug-resistant epilepsy in children from 2 to 20 years old.

The identification of the epileptogenic zone often requires making an iEEG recording for a week (implantation of intracerebral electrodes in depth).

Sometimes this recording has to be repeated, providing a unique opportunity to directly record brain activity at different periods of its development.

Children will listen to pre-recorded phrases and stories such as "The Little Prince of Antoine de Saint-Exupéry" while being recorded with iEEG.

ELIGIBILITY:
Inclusion Criteria:

* Any patient benefiting from a long-term intracranial brain recording.
* Non-opposition to participating in the study (adult patients)
* Non-opposition of at least one of the holders of the exercise of parental authority (minor patients)

Exclusion Criteria:

* Patient with complete deafness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient benefiting from a long-term intracranial brain recording
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
This is a non-clinical research study investigating from intracranial recordings how speech representation changes throughout human development. | maximum 21 days
  intracranial recordings

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique de Rothschild, Paris, France, France

IPD SHARING:
Plan to Share IPD: No